CLINICAL TRIAL: NCT04802668
Title: Factors Influencing the Reliability of Pulse Pressure Variation (PPV) as a Predictor of Fluid Responsiveness in Mechanically Ventilated Patients
Brief Title: Factors Influencing of Pulse Pressure Variation (PPV)
Acronym: FacPPV
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Clinical Professor, Southeast University, China
Other Study IDs: 20210101PPV
Record Dates: First submitted 2021-02-06; First posted 2021-03-17 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Haemodynamics; Fluid Responsiveness; Pulse Pressure Variation
Keywords: haemodynamics;; Pulse pressure variation;; fluid responsiveness;; Mechanical ventilation;

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Circulatory failure patients: Circulatory failure patients requiring fluid responsiveness evaluation
  Interventions: Device: Patients were ventilated with assist-control ventilation（A/C） mode at different tidal volume; Behavioral: spontaneous breathing and no spontaneous breathing

INTERVENTIONS:
Device: Patients were ventilated with assist-control ventilation（A/C） mode at different tidal volume — Ventilation mode was set to assist-control volume ventilation with different tidal volume, respiratory frequency 15 times/min, PEEP 5 centimeter water column.
Behavioral: spontaneous breathing and no spontaneous breathing — Data were recorded when patients had and did not have spontaneous breathing

SUMMARY:
The investigators studied the predictive value of PPV in the patients with different influencing factors;and the method to improve the predictive value,which can improve the application of PPV in ICU.

DETAILED DESCRIPTION:
PPV can be used to predict fluid responsiveness in patients with circulatory shock.However, it is affected by many factors, which leads to the decrease of the applicability of PPV in ICU.Therefore, the investigators studied the predictive value of PPV in the patients with different influencing factors;and the method to improve the predictive value,which can improve the application of PPV in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring invasive mechanical ventilation
* Acute circulatory failure,defined as:systolic blood pressure <90 mmHg or blood pressure in patients with previous hypertension lower than the baseline value> 40 mmHg; vasoactive drugs are required to maintain blood pressure (mean arterial pressure> 65 mmHg); with or without signs of hypoperfusion (oliguria<0.5ml.kg-1.h-1 for at least 2 hours; arterial blood lactic acid>2.5mmol.L-1; skin mottling)

Exclusion Criteria:

* The age of the patient is less than 18 years old or more than 80 years old
* Refuse to sign the informed consent to join the group
* Atrial fibrillation and other arrhythmias that seriously affect the output per beat;
* With pregnancy
* Other situations where the clinician believes that the patient is not suitable for inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with circulatory failure selected to enter the Department of Critical Care Medicine
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
cardiac output(CO) | 1 day
  The measurement of cardiac output(CO);

SECONDARY OUTCOMES:
measurement of Hemodynamic variables from the monitor; | 1 day
  The investigators record the hemodynamic variables from the monitor MAP and CVP
measurement of Pulse pressure variation（PPV）from monitor; | Research period
  Pulse pressure variation (PPV)(percent) ,whic is calculated from the systolic and diastolic blood pressure,can be read from the monitor directly.
measurement of airway pressure variables from ventilator | 1 day
  The investigators record the airway pressure variables during the inspiration and expiration from the ventilator
P 0.1 | 1 day
  airway occlusion pressure at 100 milliseconds after the onset of inspiration (P0.1)(cmH2O)
Pocc | 1 day
  delta change of airway pressure during expiratory occlusion in different interventions.

OTHER OUTCOMES:
Pes | 1 day
  esophageal pressure
transpulmonary pressure | 1 day
  transpulmonary pressure and delta transpulmonary pressure
Outcome | 28 day
  ICU， 28day and hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD, Study Director — professor
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chen H, Liang M, He Y, Teboul JL, Sun Q, Xie J, Yang Y, Qiu H, Liu L. Inspiratory effort impacts the accuracy of pulse pressure variations for fluid responsiveness prediction in mechanically ventilated patients with spontaneous breathing activity: a prospective cohort study. Ann Intensive Care. 2023 Aug 17;13(1):72. doi: 10.1186/s13613-023-01167-0. PMID 37592166